CLINICAL TRIAL: NCT06201338
Title: Pre-operative Screening of Functional Fragilities Before Open Aortic Surgery : a New Area
Brief Title: Pre-operative Screening of Functional Fragilities Before Open Aortic Surgery: a New Area
Acronym: Frail Aorta
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Paul Sabatier of Toulouse (Other)
Collaborators: Sarah BADICHE (Unknown)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Clinical Professor, University Paul Sabatier of Toulouse
Other Study IDs: RnIPH 2023-91
Record Dates: First submitted 2023-12-15; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Aortic Aneurysm; Aortic Occlusion
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open aortic surgery: Patient undergoing open surgery for abdominal aortic aneurysm or abdominal aortic occlusion
  Interventions: Procedure: Screening of preoperative frailty

INTERVENTIONS:
Procedure: Screening of preoperative frailty — The day before the surgery, a multimodal evaluation is performed regarding :
  Cognitive assessment: Mini mental State evaluation (MMSE) test Physical functional assessment: Chair raising Addiction assessment: Fagerstrom Assessment of the social environment: environmental assessment Nutritional assessment: Grip test Quality of life: completion of SF 36 scale and QOR15 scale

SUMMARY:
Aneurysmal or occlusive abdominal aortic pathology has seen its prevalence increase over the years despite the various cardiovascular risk factor management campaigns deployed.

Currently, a large proportion of these aortic pathologies require effective and definitive treatment by open surgery. In fact, minimally invasive endovascular treatment, which can provide good results in certain cases, cannot be generalized simply and can even lead to sometimes incomplete treatments requiring even more complex secondary open surgery.

The preoperative assessment before open aortic surgery is relatively well coded with cardiological and respiratory assessments in particular. However, the literature has so far never focused on the overall vision of the patient with a complete functional assessment which would make it possible to consider a specific preoperative fragility scale and would thus give practitioners corrective targets before such an intervention. in order to simplify the patient's post-operative journey by limiting complications.

The investigators therefore propose to collect a certain number of elements already collected in standard care in a systematic and prospective manner in order to create a risk scale. All of these elements being modifiable, they should ultimately make patients more robust for such an intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing open aortic surgery in the vascular surgery department

Exclusion Criteria:

* patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Aortic aneurysm >55mm
  * Aortic occlusion responsible for severe claudication of the lower limbs or critical ischemia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Post operative mortality | day 30 post operative
  Rate of death after surgery
Major adverse cardiovascular events (MACE) | day 30 post operative
  Rate of nonfatal stroke, nonfatal myocardial infarction and cardiovascular death
Length of stay | day 30 post operative
  Evaluation of the length of stay in days of the patients
Home discharged | day 30 post operative
  Rate of patient who need a rehabilitation center after surgery

SECONDARY OUTCOMES:
Respiratory complications | day 30 post operative
  Rate of pneumopathy and need of reintubation or intubation longer than 24h
Quality of life : 36-item Short-Form Health Survey | day 30, 3 months, 6 months, 1 year
  Evaluation of post-operative quality of life compared to pre-operative data with 36-item Short-Form Health Survey
Quality of life : Quality of Recovery-15 | day 30, 3 months, 6 months, 1 year
  Evaluation of post-operative quality of life compared to pre-operative data with Quality of life Quality of Recovery-15

CONTACTS AND LOCATIONS:
Locations (1):
- Toulouse university hospital, vascular surgery department, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided